CLINICAL TRIAL: NCT04927416
Title: The Role of 68-Gallium-DOTATATE-PET/CT in the Imaging of Metastatic Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000079; 000079-DK
Record Dates: First submitted 2021-06-15; First posted 2021-06-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-09

CONDITIONS: Metastic Thyroid Cancer
Keywords: Thyroid Cancer; Metastases; Ga68-DOTATATE; Somatostatin Receptors; Positron Emission Tomography
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Differentiated thyroid cancer (DTC) (Experimental): Patients with DTC but not HTC
  Interventions: Drug: 68-Gallium-DOTATATE-PET/CT
- Hurthle cell thyroid cancer (HTC) (Experimental): Molecularly and histologically unique subtype of DTC - Hurthle cell thyroid cancer (HTC),
  Interventions: Drug: 68-Gallium-DOTATATE-PET/CT
- Medullary thyroid cancer (MTC) (Experimental): Patients with metastatic thyroid cancer of neuroendocrine origin - medullary thyroid cancer (MTC)
  Interventions: Drug: 68-Gallium-DOTATATE-PET/CT

INTERVENTIONS:
Drug: 68-Gallium-DOTATATE-PET/CT — 68Ga-DOTATATE is administered one-time via intravenous injection of 5 mCi in a volume of 3-5 ml containing up to 50 mcg [68Ga] DOTATATE.

SUMMARY:
Background:

About 5% to 10% of differentiated thyroid cancers become resistant to standard treatment with radioactive iodine. In these cases, treatment options are limited and generally not effective. Researchers want to see if they can better detect thyroid tumors by using a compound called 68Gallium-DOTATATE. This compound may bind to a tumor and make it visible during a positron emission tomography/computed tomography (PET/CT) scan. This information might help guide future research and treatment.

Objective:

To identify the people with thyroid cancer whose tumors have a high uptake of 68Gallium-DOTATATE as analyzed by imaging with PET/CT.

Eligibility:

People ages 18 years and older with thyroid cancer that has spread outside of the thyroid.

Design:

Participants will have a medical exam. They will give blood and urine samples. Some samples will be used for research.

Participants will have imaging scans that follow standard of care. These scans may include:

CT scan of the neck, chest, abdomen, and pelvis

Bone scan

Magnetic resonance imaging of the brain, spine, or liver

18-FDG-PET/CT as needed

Participants will have a PET/CT scan. They will get an intravenous (IV) line. They will get an IV injection of 68Gallium-DOTATATE. It contains radioactive tracers. The PET/CT scanner is shaped like a large donut. It contains crystals. The crystals pick up small radiation signals that are given off by the tracers. The CT part of the scan uses low-dose x-rays. The pictures made by the scanner show where the tracers are in the body. The session will last 90 minutes.

Participation will last for about 3 months....

DETAILED DESCRIPTION:
Study Description:

The study is designed to identify the patients with metastatic radioactive iodine (RAI) non-avid or non-responsive thyroid cancer, whose tumors are characterized by the high expression of somatostatin receptors type 2 (SSTR2) by imaging with 68Gallium(68Ga)-DOTATATE Positron Emission Tomography/Computed Tomography (PET/CT). Participants will undergo a one-time experimental imaging with 68Ga-DOTATATE PET/CT. This imaging will enable identification of patients with high maximum standard uptake value (SUVmax) of 68Ga-DOTATATE defined as SUVmax of >15, as this SUVmax threshold has been associated with a good response to peptide receptor radionuclide therapy (PRRT) in pre-clinical and clinical models of SSTR2-positive tumors. PRRT will not be offered in this trial.

Objectives:

Primary Objective:

To compare the prevalence of patients with metastatic RAI-non-avid or RAI-non-responsive thyroid cancer whose tumors are characterized by a high SSTR2 expression by imaging with 68Ga-DOTATATE PET/CT between three groups:

* Group HTC--the molecularly and histologically unique subtype of differentiated thyroid cancer (DTC) - Hurthle cell thyroid cancer (HTC),
* Group DTC--patients with remaining histological types of DTC,
* Group MTC--patients with metastatic thyroid cancer of neuroendocrine origin - medullary thyroid cancer (MTC).

Secondary Objectives:

1. To analyze the association between the 68Ga-DOTATATE uptake and molecular signature of thyroid cancer and tumor volume,
2. to create a repository of data for future research in thyroid cancer.

Endpoints:

Primary Endpoint: Prevalence of thyroid cancer patients characterized by a high SSTR2 expression in at least one metastatic lesions per patient documented by SUVmax of 68Ga-DOTATATEPET/CT of above 15 among patients with metastatic HTC, DTC and MTC.

Secondary Endpoints: Associations between 68Ga-DOTATATE uptake as measured by SUVmax in up to 10 lesions per organ per patient and:

1. Somatic mutation status in primary tumors divided into BRAF-like, RAS-like, harboring mitochondrial DNA mutations and /or RET protooncogene mutation,
2. Tumor volume measured in cm3 per the ellipsoid formula p/6 length*width*depth.

ELIGIBILITY:
* INCLUSION CRITERIA:

Data prospectively collected from the 28 subjects enrolled under this protocol, and data from 26 subjects collected under 77-DK-0096 and/or 00-CH-0093 will be analyzed. Among the 26 subjects prospectively evaluated under 77-DK-0096 protocol, 21 out of 26 had research 68Ga-DOTATATE PET/CT performed under the DOTATATE sub-study of 77-DK-0096, and 5 out of 26 had 68Ga-DOTATATE PET/CT done under 00-CH-0093. Again, the inclusion of the above data was per the IRB s request to transition the sub-study into a new standalone protocol. This will give us a total of 54 subjects for the final analyses, with at least 18 subjects from each group (e.g., HTC, DTC, and MTC), which is required to meet the primary objectives of this study with sufficient power of 80% and type 1 error alpha of < 0.05.

Patients with HTC, DTC, and MTC will be identified by the investigators. The potential candidates for the study will be screened for eligibility to participate in the study and invited to sign the Research 68Ga-DOTATATE PET/CT imaging informed consent form. The same inclusion/exclusion criteria were applied to the subjects who underwent imaging with the 68GADOTATATE PET/CT, either under the 77-DK-0096 sub-study or as clinically-indicated imaging under 00-CH-0093.

In order to be eligible to participate in this study, an individual with DTC (including HTC) must meet all of the following criteria:

* Male or female, aged >18 years.
* Patients with established thyroid cancer diagnosis presenting with either:

  * Locally advanced or distant metastases, which are RAI-non-avid based on the or diagnostic or post-treatment whole body scan (WBS)

OR

--Patients with RAI-non-responsive disease, who have the evidence of disease progression defined by RECIST 1.1 criteria after therapy with RAI.

In order to be eligible to participate in this study, an individual with MTC must meet all of the following criteria:

* Male or female, aged >18 years.
* Patients with locally advanced or metastatic MTC or patients suspected of locally advanced or metastatic MTC with calcitonin level > 500 pg/mL.

EXCLUSION CRITERIA:

Subjects with either HTC, DTC, or MTC who meet any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation by self-report.
* Serious underlying medical conditions that restrict diagnostic testing or therapy such as renal failure, congestive cardiac failure or active coexisting non-thyroid carcinoma;
* Patients unable to give informed consent.

Ages: 18 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with metastatic RAI-non-avid or RAI-non-responsive thyroid cancer whose tumors are characterized by a high SSTR2 expression by imaging with 68Ga-DOTATATE PET/CT | During baseline assessment
  Prevalence of thyroid cancer patients characterized by a high SSTR2 expression in at least one metastatic lesion per patient documented by SUVmax of 68Ga-DOTATATE-PET/CT of above 15 among patients with metastatic HTC, DTC and MTC.

SECONDARY OUTCOMES:
Correlation between tumor volume and SUV max for each participant | During baseline assessment
  Tumor volume in cm3 as measured by the ellipsoid formula will be measured on up to 10 lesions per organ and correlated with SUVMax
Maximum standard uptake value (SUVmax) of 68Ga-DOTATATE | During baseline assessment
  SUVmax will be compared in groups based on the somatic mutation status in primary tumors: BRAF-like, RAS-like, harboring mitochondrial DNA mutations and /or RET protooncogene mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000079-DK.html